CLINICAL TRIAL: NCT06498284
Title: HM-002-1005 - A Phase 1, Randomized, Double Blind, Placebo Controlled, Single Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Subjects With Type 2 Diabetes Mellitus
Brief Title: Evaluate HM-002-1005 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMM0125
Record Dates: First submitted 2024-04-30; First posted 2024-07-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Glucokinase agonist; HM-002-1005; Hyperglycemia; Diabetes Mellitus, Type II; Single dose escalation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: single oral dose escalation study
Who Masked: Participant, Investigator
Masking Description: matching placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HM-002-1005 61.5 mg or matching placebo (Experimental): Single dose of 61.5 mg HM-002-1005 or matching placebo
  Interventions: Drug: HM-002-1005
- HM-002-1005 123 mg or matching placebo (Experimental): Single dose of 123 mg HM-002-1005 or matching placebo
  Interventions: Drug: HM-002-1005
- HM-002-1005 184.5 or 246 mg, or matching placebo (Experimental): Single dose of 184.5 or 246 mg HM-002-1005 or matching placebo
  Interventions: Drug: HM-002-1005
- HM-002-1005 369 mg or matching placebo (Experimental): Single dose of 369 mg HM-002-1005 or matching placebo
  Interventions: Drug: HM-002-1005

INTERVENTIONS:
Drug: HM-002-1005 — HM-002-1005 extended release tablets for oral administration compared with matching placebo tablets
  Other Names: 1005

SUMMARY:
The purposes of this study are to:

* Evaluate the safety and tolerability of the study drug.
* Measure how much of the study drug (HM-002-1005) and its breakdown product get into the bloodstream, and how long it takes the body to get rid of them.
* Measure the amount of glucose (blood sugar) and a substance called C-peptide in the bloodstream after receiving the study drug.

Researchers will compare the study drug to a placebo (a look-alike substance that contains no drug).

Participants will:

* Stay 5 days and 4 nights or 6 days and 5 nights at the research site, and have a follow-up phone call 7 days after leaving the research site.
* Take one (1) dose of the study drug or placebo
* Have blood taken to measure the amount of study drug and its breakdown product and the levels of glucose and C-peptide
* Have safety tests such as vital sign, ECGs, and glucose measurements

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 65 years of age, inclusive.
2. Body mass index between 18.5 and 38.0 kg/m2, inclusive.
3. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
4. Type 2 diabetes mellitus, as determined by the American Diabetes Association (ADA) Standard Care Diagnostic Criteria 2023, and

   1. are drug naïve, treated with diet and exercise, or
   2. have been on a stable dose of ≤2000 mg metformin for ≥1 month, or
   3. have been on a stable dose of antidiabetic medications (other than metformin) for ≥90 days.
5. Except for findings consistent with T2DM, in good health, determined from medical history, 12 lead electrocardiogram (ECG), vital signs measurements, clinical laboratory evaluations, and physical examinations at screening and/or check in, as assessed by the investigator (or designee).
6. Glycated hemoglobin between 6.5% and 9.5%, inclusive.
7. Fasting plasma glucose between 126 and 196 mg/dL (7 and 11 mmol/L, respectively), inclusive. Testing may be repeated once, at the discretion of the investigator (or designee).

   Other Inclusions
8. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

1. Type 1 diabetes mellitus, maturity onset diabetes of the young, or diabetes mellitus caused by damage to the pancreas or any other condition (eg, acromegaly or Cushing's syndrome).
2. Diabetic neuropathy, retinopathy, or nephropathy.
3. Acute or chronic metabolic acidosis, including diabetic ketoacidosis.
4. History of severe hypoglycemia, defined as severe cognitive impairment requiring external assistance for recovery within 3 months prior to dosing; or recurrent hypoglycemia (Level 2), defined as ≥2 episodes within 3 months prior to dosing; or ADA Level 3 hypoglycemia within 6 months prior to dosing.
5. Hypoglycemia unawareness or asymptomatic hypoglycemia.
6. Clinically significant history of liver disease (eg, hepatitis and cirrhosis) within 1 year prior to screening.
7. Clinically significant history of renal disease. Mild to moderate chronic kidney disease is permitted.
8. Clinically significant history of cardiovascular disease, particularly coronary artery disease, arrhythmias, atrial tachycardia, or congestive heart disease within 1 year prior to screening. Managed hypertension is permitted.
9. Clinically significant history of any central nervous system disease, including transient ischemic attack, stroke, seizure disorder, depression, or behavioral disturbances within 1 year prior to screening.
10. Clinically significant gastric emptying abnormality (eg, severe diabetic gastroparesis or gastric outlet obstruction) or have had gastric bypass surgery.
11. Clinically significant or unstable history of any hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
12. Known or active malignancy, except basal cell carcinoma and cutaneous squamous cell carcinoma.
13. Any hospital admission or major surgery within 90 days prior to screening.
14. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, as determined by the investigator (or designee).
15. Fasting C peptide <0.81 ng/mL.
16. Alanine aminotransferase, aspartate aminotransferase, or gamma glutamyl transferase >2 × the upper limit of normal (ULN); or total bilirubin >1.5× ULN.
17. Uncontrolled hypertriglyceridemia >500 mg/dL.
18. Estimated glomerular filtration rate ≤45 mL/min/1.73 m2, as calculated using the 2021 Chronic Kidney Disease Epidemiology equation.
19. QT interval corrected for heart rate using Fridericia's method >450 msec.
20. Positive hepatitis panel and/or positive human immunodeficiency virus test .
21. Positive pregnancy test.
22. Use of insulin, sulfonylureas, and glinides (eg, repaglinide and nateglinide).
23. Use of any strong or moderate cytochrome P450 (CYP) 3A4 inducers within 28 days prior to dosing or any strong or moderate CYP3A4 inhibitors within 7 days or 5 half lives, whichever is longer, prior to dosing.
24. Use of any P glycoprotein inducers within 14 days prior to dosing or any P glycoprotein inhibitors within 5 days or 5 half lives, whichever is longer, prior to dosing
25. Use of any carboxylesterase 2 inhibitors within 5 days or 5 half lives, whichever is longer, prior to dosing Note: The use of hypertensive therapies is permitted, providing that they are do not meet exclusion criteria 22 to 25.
26. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days.
27. Positive alcohol test result, or positive urine drug screen (confirmed by repeat), or positive cotinine test at screening or check in.
28. Current drug abuse, defined as the use of any illegal substance or misuse or excessive used of over the counter or prescription drugs; or current alcohol abuse, defined as the inability to stop or control alcohol use, despite adverse social or health consequences.
29. Consumption of alcohol, or caffeine containing foods or beverages within 48 hours, or foods and beverages containing grapefruit or Seville oranges within 7 days prior to check in.
30. Use of tobacco or nicotine containing products within 6 months prior to check in.
31. Receipt or donation of >1 unit (approximately 450 mL) of blood products within 3 months prior to screening.
32. Poor peripheral venous access.
33. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 11 Days
  incidence and severity of adverse events from Day1 to Day 11
Area under the plasma concentration versus time curve (AUC) | 72 hour
  area under the concentration-time curve from time 0 to 72 hours postdose of HM-002-1005 in plasma
maximum observed concentration (Cmax) | 72 hours
  Cmax of HM-002-1005 in plasma
time of the maximum observed concentration (Tmax) | 72 hours
  Tmax of HM-002-1005 in plasma
apparent terminal elimination half life (t1/2) | 72 hours
  t1/2 of HM-002-1005 in plasma

SECONDARY OUTCOMES:
glucose concentration following single oral dose of HM-002-1005 | 24 hours
  serum glucose concentration over 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Prezioso, MD, Principal Investigator — Clinical Pharmacology of Miami
Locations (1):
- Clinical Pharmacology of Miami, Hialeah, Florida, United States